CLINICAL TRIAL: NCT02647866
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled Multiple Ascending Dose Study (Induction Therapy) & Long-term Extension Therapy of an Anti-OX40 Monoclonal Antibody (KHK4083) in Subjects With Moderately Active UC
Brief Title: Study of a Monoclonal Antibody KHK4083 in Moderate Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin, Inc. (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4083-002
Record Dates: First submitted 2015-12-08; First posted 2016-01-06 (Estimated); Results first posted 2020-03-05 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Ulcerative Colitis; Digestive System Diseases; Colitis, Ulcerative; Colitis; Gastrointestinal Diseases; Inflammatory Bowel Diseases; Intestinal Diseases; Colonic Diseases; Autoimmune Disease; Abdominal Pain
Keywords: 4083-002; Intestinal Diseases; Ulcerative Colitis; UC; Mayo Clinic Scoring; Gastrointestinal Tract
MeSH Terms: conditions — Colitis, Ulcerative; Digestive System Diseases; Colitis; Gastrointestinal Diseases; Inflammatory Bowel Diseases; Intestinal Diseases; Colonic Diseases; Autoimmune Diseases; Abdominal Pain | interventions — KHK4083

STUDY DESIGN:
Intervention Model Description: Double-blind Induction Therapy was separated into Part A for administration of multiple ascending IV doses of KHK4083 (or placebo) to subjects in Cohorts 1-3 and Part B for administration of the maximally tolerated dose (as determined in cohorts 1-3) in expansion cohort 4. Subjects in Part A were prohibited from participating in Part B.
  Subjects in each cohort were randomly assigned in a 3:1 ratio to receive KHK4083 or placebo by IV infusion over 60 minutes (± 10 min.). Each subject received a total of 6 treatments (1 IV infusion per treatment) every 2 weeks from Week 0 (Day 1) to Week 10.
  Subjects who completed double-blind Induction Therapy (i.e., at least 5 of 6 treatments) and had a clinical response or mucosal healing, as defined above, were eligible to continue in double-blind Long Term Extension Therapy (Weeks 12-52) & after protocol amendment all subjects who received at least 5 of 6 treatments were eligible for Open Label Extension Therapy (Weeks 12-52).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- KHK4083 Cohort 1 (Experimental): Subjects received one 1.0 mg/kg IV infusion treatment of KHK4083 every two weeks from Week 0 to Week 10 of Induction Therapy. Subjects who chose to continue into extension therapy and were eligible received one IV infusion every 4 weeks (at the same dose as Induction Therapy) from Week 12 to Week 48.
  Interventions: Drug: KHK4083
- KHK4083 Cohort 2 (Experimental): Subjects received one 3.0 mg/kg IV infusion treatment of KHK4083 every two weeks from Week 0 to Week 10 of Induction Therapy. Subjects who chose to continue into extension therapy and were eligible received one IV infusion every 4 weeks (at the same dose as Induction Therapy) from Week 12 to Week 48.
  Interventions: Drug: KHK4083
- KHK4083 Cohort 3 (Experimental): Subjects received one 10.0 mg/kg IV infusion treatment of KHK4083 every two weeks from Week 0 to Week 10 of Induction Therapy. Subjects who chose to continue into extension therapy and were eligible received one IV infusion every 4 weeks (at the same dose as Induction Therapy) from Week 12 to Week 48.
  Interventions: Drug: KHK4083
- KHK4083 Cohort 4 (Experimental): Subjects received one maximum tolerated dose (10.0 mg/kg) IV infusion treatment of KHK4083 every two weeks from Week 0 to Week 10 of Induction Therapy. Subjects who chose to continue into extension therapy and were eligible received one IV infusion every 4 weeks (at the same dose as Induction Therapy) from Week 12 to Week 48.
  Interventions: Drug: KHK4083
- Placebo (Placebo Comparator): Subjects received one IV infusion treatment of Placebo every two weeks from Week 0 to Week 10 of Induction Therapy. Subjects who chose to continue into extension therapy and were eligible received one IV infusion every 4 weeks (at the same dose as Induction Therapy) from Week 12 to Week 48. Subjects who participated in Open-Label Therapy received KHK4083 instead of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KHK4083 — IV Infusion
  Arms: KHK4083 Cohort 1; KHK4083 Cohort 2; KHK4083 Cohort 3; KHK4083 Cohort 4
Drug: Placebo — IV Infusion
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety and tolerability of administration of multiple ascending doses of KHK4083 and to select the highest dose tolerated by subjects with moderately active Ulcerative Colitis (UC) followed by a Long-term Extension Therapy (LTE) phase for eligible subjects with a clinical response.

DETAILED DESCRIPTION:
A Phase 2, double-blind clinical study of multiple ascending doses of KHK4083 (or placebo) with an Long-term Extension Therapy (LTE) phase will be conducted in approximately 60 randomized adult subjects with moderately active UC who have a documented unsuccessful previous treatment.

The Treatment Period includes double-blind Induction Therapy (12 weeks) and Open-label Therapy (OLE) phase (40 weeks) for eligible subjects at Week 12. Subjects already enrolled in the double-blind, long-term extension (LTE) under preceding versions of the protocol who worsen may be eligible to transition to the OLE up to Week 28.

The Follow Up Period after the last administration will be for up to 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is able and willing to comply with study procedures, and to adhere to dosing, visit schedules and follow-up procedures as described in the protocol and ICF;
2. Subject voluntarily signs/dates an Institutional Review Board (IRB)/Independent Ethics Committee (IEC)-approved ICF in accordance with regulatory and Institutional Guidelines;
3. Male and female subjects ≥ 18 years of age at the time of enrollment;
4. Subject has UC that was diagnosed at least 6 months prior to the Screening visit;
5. Subject has moderately active UC with a total Mayo score of 4-9 and an endoscopic sub-score of at least 2, with disease that extends at least 15 cm from the anal verge;
6. Subject has had previous treatment (within 5 years prior to Screening) with one or more of the following: corticosteroids, immunosuppressive medications or TNF antagonist therapy that was unsuccessful because of a lack of efficacy response.
7. Female subjects (WOCBP) must have a negative pregnancy test at Screening and Baseline. WOCBP must agree to use effective contraception;
8. Male subjects (including those who have had a vasectomy) must use adequate contraception during the study and for at least 6 months after the last dose of investigational product.

Exclusion Criteria:

1. Subject, who, for any reason, is judged by the Investigator to be inappropriate for this study;
2. Subject has a medical history of other clinically significant diseases/disorders;
3. Two or more biologic treatments with different mechanisms of action (e.g., infliximab, vedolizumab and golimumab) or Three or more anti-TNF biologics e.g. infliximab, adalimumab
4. Subject requires prescription treatment for UC, except for the stable, oral treatment of UC for 4 weeks prior to screening.
5. Subject has received any of the following prior treatments or treatments within the specified time prior to the Baseline visit:

   * Natalizumab, efalizumab, rituximab or other lymphocyte-depleting treatments, including but not limited, to alkylating agents (such as cyclophosphamide or chlorambucil) and total lymphoid irradiation at any time;
   * TNF antagonists within 8 weeks, or 5 half-lives (up to 12 weeks);
   * Vedolizumab within 16 weeks;
   * Methotrexate, cyclosporine, mycophenolate, tacrolimus, thalidomide, or other immune altering drugs within 4 weeks (ophthalmologic preparations are permitted);
   * 5-ASA enema, steroid enema or suppository use within 2 weeks ; and/or Investigational agents within 8 weeks or 5 half-lives (whichever is longer).
6. Subject with recent, suspected or confirmed symptomatic stenosis of the colon, abdominal abscess, or ischemic colitis based on clinical or radiographic data; a history of toxic megacolon; or who had any previous surgery for UC;
7. Subject with known colonic dysplasia, adenomas or polyposis;
8. Subject had major surgery within 4 weeks prior to Screening or an anticipated requirement for major surgery;
9. Subject with enteric pathogens (including Clostridium difficile);
10. Subject with any of the following hematological and chemistry laboratory values:

    * Platelet count < 100,000/mm3;
    * Neutrophils < 1500/mm3;
    * Serum creatinine ≥ 1.6 mg/dL (≥ 144.4 μmol/L);
    * Alkaline phosphatase > 3 times the upper limit of normal (ULN);
    * AST or ALT > 2 times ULN;
    * Total bilirubin > 2 mg/dL, unless due to Gilbert's Syndrome;
    * Serum albumin < 3 g/dL;
    * Hemoglobin < 9 g/dL;
    * Glycated serum hemoglobin A1c ≥ 9%.
11. Subject has clinically significant cardiac disease;
12. Subject is pregnant or breastfeeding;
13. Subject has had major immunologic reaction;
14. Subject is Hepatitis B core antibody or surface antigen positive and/or Hepatitis C antibody positive with detectable RNA;
15. Subject has a history of human immunodeficiency virus (HIV) positivity, tests positive for HIV, or has congenital or acquired immunodeficiency;
16. Subject has or has had active TB, suspected extra-pulmonary TB, a history of incompletely treated TB, or latent TB or other latent infection. Subjects with latent TB (clinical findings, purified protein derivative [PPD] or interferon gamma release assay [IGRA]) may be included in the study if prophylactic therapy for latent TB is started at least 4 weeks prior to Screening. Subjects with a potentially untreated other infection (clinical findings) are to be excluded.
17. Subject has bacterial infections requiring treatment with oral or parenteral antibiotics, within 2 and 4 weeks, respectively.
18. Subject has a history of systemic opportunistic infection or recurrent infections
19. Subject has malignancy or history of malignancy, except for adequately treated basal cell skin cancer or adequately treated carcinoma in-situ of the cervix without recurrence at least 5 years.
20. Subject who received a bacille Calmette-Guérin (BCG) vaccine within 6 months of randomization or live vaccination (e.g., measles, mumps, rubella [MMR]; herpes zoster; varicella, intranasal influenza; and oral poliomyelitis) within 4 weeks of randomization.
21. Subject with a history of or active substance abuse.
22. Subject has other severe acute or chronic medical or psychiatric condition or laboratory abnormality.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Strout, MBA, Study Director — Kyowa Kirin, Inc.
Locations (18):
- Greenville, South Carolina, United States
- Czechia (2):
  - Hradec Králové
  - Znojmo
- Budapest, Hungary
- Poland (5):
  - Bydgoszcz
  - Rzeszów
  - Sopot
  - Tychy
  - Warsaw
- Bucharest, Sector 2, Romania
- Russia (5):
  - Krasnoyarsk
  - Moscow
  - Novosibirsk
  - Penza
  - Saint Petersburg
- Serbia (3):
  - Zemun, Belgrade
  - Bežanija Kosa, Belgrade
  - Kragujevac

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Investigative sites in the US, Poland, Czech Republic, Russia, Romania, Serbia, and Hungary screened patients from January 2016 until June 2017, with the first patient enrolled in June 2016.
Pre-assignment Details: A total of 109 patients were screened during the recruiting period. Subjects were enrolled into the study only if all inclusion criteria and none of the exclusion criteria were fulfilled.
Period: Overall Study
Arm/Group | KHK4083 Cohort 1 | KHK4083 Cohort 2 | KHK4083 Cohort 3 | KHK4083 Cohort 4 | Placebo
Started | 9 | 10 | 9 | 21 | 17
Completed Induction Therapy | 8 (Subjects received KHK4083 1.0 mg/kg for 12 weeks) | 9 (Subjects received KHK4083 3.0 mg/kg for 12 weeks) | 8 (Subjects received KHK4083 10.0 mg/kg for 12 weeks) | 19 (Subjects received the maximum tolerated dose of KHK4083 10.0 mg/kg for 12 weeks) | 17 (Subjects received Placebo for 12 weeks)
Completed Induction Therapy Follow-Up | 5 | 1 | 2 | 0 | 2
Completed Long-Term Extension Therapy | 3 (10 add'l treatments of KHK4083 (same dose as Induction Therapy) as maintenance therapy.) | 0 | 0 | 0 | 0
Completed LTE Follow-up | 2 | 0 | 0 | 0 | 0
Completed Open-Label Extension Therapy | 0 | 7 (10 add'l treatments of Open-Label KHK4083 (same dose as Induction Therapy) as maintenance therapy.) | 4 (10 add'l treatments of Open-Label KHK4083 (same dose as Induction Therapy) as maintenance therapy) | 17 (10 add'l treatments of Open-Label KHK4083 (same dose as Induction Therapy) as maintenance therapy) | 13 (10 add'l treatments of Open-Label KHK4083 (same dose as Induction Therapy) as maintenance therapy)
Completed OLE Follow-up | 0 | 6 | 4 | 14 | 10
Moved From LTE to OLE Therapy | 0 | 5 | 0 | 0 | 2
Discontinued the Treatment | 4 | 5 | 5 | 5 | 8
Discontinued the Study | 5 | 4 | 5 | 6 | 8
Completed | 4 | 6 | 4 | 15 | 9
Not Completed | 5 | 4 | 5 | 6 | 8
Not completed — Adverse Event | 0 | 0 | 2 | 2 | 1
Not completed — Disease Worsening | 3 | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 2 | 4 | 4
Not completed — Physician Decision | 0 | 1 | 1 | 0 | 2
Not completed — Death | 0 | 1 | 0 | 0 | 0
Not completed — Subject moved to different country | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | KHK4083 Cohort 1 | KHK4083 Cohort 2 | KHK4083 Cohort 3 | KHK4083 Cohort 4 | Placebo | Total
Number analyzed (Participants) | 9 | 10 | 9 | 21 | 17 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 8 | 9 | 19 | 17 | 60
  >=65 years | 2 | 2 | 0 | 2 | 0 | 6
Age, Continuous [Mean (Full Range); unit: years] | 47.3 [18 to 67] | 46.1 [21 to 75] | 41.2 [18 to 63] | 41.1 [18 to 78] | 33.8 [18 to 61] | 40.8 [18 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 5 | 6 | 8 | 25
  Male | 5 | 8 | 4 | 15 | 9 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 10 | 9 | 21 | 17 | 66
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 1
  White | 9 | 10 | 9 | 21 | 16 | 65
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Treatment-related Adverse Events
Description: To determine the safety and tolerability of KHK4083
Time Frame: Up to 52 weeks
Population: Safety Analysis Set - All randomized subjects who received any (even partial dose) investigational product (KHK4083 or placebo).
Measure: Count of Participants; unit: Participants
Groups:
- KHK4083 Combined: The total number of participants analyzed who were randomized to KHK4083 during Induction Therapy.
- Placebo: Subjects received placebo IV infusion treatments from Baseline to Week 12. Subjects who completed double-blind Induction Therapy (i.e., at least five of six treatments) were eligible to enter OLE Therapy and receive 10 treatments of open-label KHK4083 (at the same dose administered to that subject during Induction Therapy) as maintenance therapy. Each subject was to receive one IV infusion every 4 weeks from Week 12 to Week 48.
Arm/Group | KHK4083 Cohort 1 | KHK4083 Cohort 2 | KHK4083 Cohort 3 | KHK4083 Cohort 4 | KHK4083 Combined | Placebo
Number analyzed (Participants) | 9 | 10 | 9 | 21 | 49 | 17
Participants
  With Any TEAE | 5 | 7 | 7 | 14 | 33 | 13
  With Any Drug-related TEAE | 3 | 2 | 3 | 3 | 11 | 2
  With Any TEAE with an Outcome of Death | 0 | 1 | 0 | 0 | 1 | 0

2. Primary Outcome: Number of Subjects With Treatment-related Serious Adverse Events
Description: To determine the safety and tolerability of KHK4083
Time Frame: Up to 52 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- KHK4083 Combined: The total number of participants analyzed who received KHK4083 during Induction Therapy.
Arm/Group | KHK4083 Cohort 1 | KHK4083 Cohort 2 | KHK4083 Cohort 3 | KHK4083 Cohort 4 | KHK4083 Combined | Placebo
Number analyzed (Participants) | 9 | 10 | 9 | 21 | 49 | 17
Participants
  With Any Serious TEAE | 1 | 1 | 1 | 3 | 6 | 3
  With Any Drug-related Serious TEAE | 0 | 0 | 0 | 0 | 0 | 0
  Who Died | 0 | 1 | 0 | 0 | 1 | 0

3. Primary Outcome: Number of Subjects Who Show Improvement in the Mucosa at Week 12
Description: Measured by the modified Mayo endoscopy sub-score (mMES), which ranges from 0-3 with higher scores = more severe disease.
Time Frame: 12 weeks
Population: Full analysis set - All randomized subjects who received at least one full dose of investigational product and had a Baseline and at least one post-treatment primary efficacy variable.
Measure: Count of Participants; unit: Participants
Groups:
- KHK4083 Cohorts 3 + 4 Combined: Subjects received one 10.0 mg/kg IV infusion treatment of KHK4083 every two weeks from Week 0 to Week 10 of Induction Therapy. Subjects who chose to continue into extension therapy and were eligible received one IV infusion every 4 weeks (at the same dose as Induction Therapy) from Week 12 to Week 48.
Arm/Group | KHK4083 Cohort 1 | KHK4083 Cohort 2 | KHK4083 Cohorts 3 + 4 Combined | KHK4083 Combined | Placebo
Number analyzed (Participants) | 7 | 8 | 22 | 37 | 15
Participants
  mMES Improvement | 2 | 4 | 9 | 15 | 5
  Modified Baron Endoscopic Score Improvement | 3 | 5 | 8 | 16 | 6

4. Primary Outcome: Proportion of Subjects Who Show Improvement in the Mucosa at Week 52
Description: as for outcome 3
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Groups:
- KHK4083 Combined: The total number of participants analyzed who were randomized to KHK4083 during Induction Therapy,
Arm/Group | KHK4083 Cohort 1 | KHK4083 Cohort 2 | KHK4083 Cohorts 3 + 4 Combined | KHK4083 Combined | Placebo
Number analyzed (Participants) | 7 | 8 | 21 | 36 | 14
Participants | 1 | 3 | 9 | 13 | 4

5. Secondary Outcome: Number of Subjects With Confirmed Anti-KHK4083 Antibodies (Immunogenicity)
Description: The immunogenicity was assessed by determination of the development of anti-drug antibodies (ADA) against KHK4083.
Time Frame: 52 weeks
Population: All subjects who received at least one dose of KHK4083, including 14 subjects initially randomized to placebo and who then continued into Open-Label Extension therapy, where they received the maximum tolerated dose of KHK4083.
Measure: Count of Participants; unit: Participants
Arm/Group | KHK4083 Cohort 1 | KHK4083 Cohort 2 | KHK4083 Cohort 3 | KHK4083 Cohort 4 | Placebo
Number analyzed (Participants) | 9 | 10 | 9 | 21 | 14
Participants
  Subjects with Pre-Existing ADA at Baseline | 1 | 2 | 1 | 0 | 1
  Subjects with Production of Treatment-Induced ADA | 3 | 0 | 1 | 5 | 4

6. Secondary Outcome: Number of Subjects Who Achieve Mucosal Healing at Week 12
Description: The endoscopic Mayo Score (Mayo endoscopic subscore) evaluates ulcerative colitis stage, based only on endoscopic exploration. The scale ranges from 0 to 3, with higher scores = more severe activity. Mucosal healing is defined as modified Mayo endoscopy sub-score (mMES) of 0 or 1 at Week 12.
Time Frame: 12 weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | KHK4083 Cohort 1 | KHK4083 Cohort 2 | KHK4083 Cohorts 3 + 4 Combined | KHK4083 Combined | Placebo
Number analyzed (Participants) | 7 | 8 | 22 | 37 | 15
Participants | 1 | 3 | 8 | 12 | 4

7. Secondary Outcome: Number of Subjects Who Achieve Mucosal Healing at Week 52
Description: The endoscopic Mayo Score (Mayo endoscopic subscore) evaluates ulcerative colitis stage, based only on endoscopic exploration. The scale ranges from 0 to 3, with higher scores = more severe activity. Mucosal healing is defined as modified Mayo endoscopy sub-score (mMES) of 0 or 1.
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | KHK4083 Cohort 1 | KHK4083 Cohort 2 | KHK4083 Cohorts 3 + 4 Combined | KHK4083 Combined | Placebo
Number analyzed (Participants) | 7 | 8 | 21 | 36 | 14
Participants | 1 | 3 | 7 | 11 | 3

8. Secondary Outcome: Number of Subjects Who Achieve Clinical Improvement at Week 12
Description: The Mayo Clinic Score is comprised of 4 parts: stool frequency, rectal bleeding, endoscopic findings and physician's global assessment, each scored from 0-3. The total score ranges from 0-12 with higher scores indicating increased severity of disease. Improvement will be based on a reduction in the total Mayo Clinic score.
Time Frame: 12 weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | KHK4083 Cohort 1 | KHK4083 Cohort 2 | KHK4083 Cohorts 3 + 4 Combined | KHK4083 Combined | Placebo
Number analyzed (Participants) | 7 | 8 | 22 | 37 | 15
Participants | 2 | 4 | 9 | 15 | 5

9. Secondary Outcome: Change From Baseline in Total Mayo Scale Score at Week 52
Description: The Mayo Clinic Score is comprised of 4 parts: stool frequency, rectal bleeding, endoscopic findings and physician's global assessment, each scored from 0-3. The total score ranges from 0-12 with higher scores indicating increased severity of disease. Improvement was based on a reduction (mean change from Baseline [Week 0] to Week 52) in the total Mayo Clinic score.
Time Frame: 52 weeks
Population: The overall number of participants is the number in the full analysis set. The number of patients analyzed is the number of patients who had values at the noted visits.
  There were no subjects in the 10.0 mg/kg KHK4083 group in the LTE Therapy Period. There were no subjects in the 1.0 mg/kg KHK4083 group in the OLE Therapy Period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KHK4083 Cohort 1 | KHK4083 Cohort 2 | KHK4083 Cohorts 3 + 4 Combined | KHK4083 Combined | Placebo
Number analyzed (Participants) | 7 | 8 | 22 | 37 | 15
score on a scale
  LTE Period - Baseline Score: number analyzed (Participants) | 3 | 5 | 0 | 8 | 2
  LTE Period - Baseline Score | 8.0 (0.0) | 7.8 (0.8) |  | 7.9 (0.6) | 7.5 (2.1)
  LTE Period - Week 52 Score: number analyzed (Participants) | 2 | 0 | 0 | 2 | 0
  LTE Period - Week 52 Score | 2.5 (2.1) |  |  | 2.5 (2.1) |
  LTE Period - Week 52 Change from Baseline: number analyzed (Participants) | 2 | 0 | 0 | 2 | 0
  LTE Period - Week 52 Change from Baseline | -5.5 (2.1) |  |  | -5.5 (2.1) |
  OLE Period - Baseline Score: number analyzed (Participants) | 0 | 8 | 21 | 29 | 14
  OLE Period - Baseline Score |  | 7.6 (1.1) | 7.8 (1.5) | 7.8 (1.4) | 7.6 (0.9)
  OLE Period - Week 52 Score: number analyzed (Participants) | 0 | 6 | 19 | 25 | 8
  OLE Period - Week 52 Score |  | 3.7 (3.1) | 3.6 (2.4) | 3.6 (2.5) | 4.3 (3.4)
  OLE Period - Week 52 Change from Baseline: number analyzed (Participants) | 0 | 6 | 19 | 25 | 8
  OLE Period - Week 52 Change from Baseline |  | -4.0 (2.4) | -4.4 (2.7) | -4.3 (2.5) | -3.5 (2.8)

10. Secondary Outcome: Number of Subjects Who Achieve a Clinical Response at Week 12
Description: The Mayo Clinic Score is comprised of 4 parts: stool frequency, rectal bleeding, endoscopic findings and physician's global assessment, each scored from 0-3. The total score ranges from 0-12 with higher scores indicating increased severity of disease. Clinical Response is a reduction in the total Mayo Clinic score of at least 3 points.
Time Frame: 12 weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | KHK4083 Cohort 1 | KHK4083 Cohort 2 | KHK4083 Cohorts 3 + 4 Combined | KHK4083 Combined | Placebo
Number analyzed (Participants) | 7 | 8 | 22 | 37 | 15
Participants | 3 | 8 | 11 | 22 | 9

11. Secondary Outcome: Number of Subjects Who Achieve a Clinical Response at Week 52
Description: The Mayo Clinic Score is comprised of 4 parts: stool frequency, rectal bleeding, endoscopic findings and physician's global assessment, each scored from 0-3. The total score ranges from 0-12 with higher scores indicating increased severity of disease. Clinical Response indicates the change from Baseline in the Total Mayo Clinic score <= -3 and the percentage change from Baseline in the Total Mayo Clinic score <= -30% to Week 12, with an accompanying decrease in the rectal bleeding subscore of at least 1 point or an absolute rectal bleeding subscore of <= 1.
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | KHK4083 Cohort 1 | KHK4083 Cohort 2 | KHK4083 Cohorts 3 + 4 Combined | KHK4083 Combined | Placebo
Number analyzed (Participants) | 7 | 8 | 21 | 36 | 14
Participants | 2 | 4 | 14 | 20 | 5

12. Secondary Outcome: Number of Subjects Who Achieve Clinical Remission at Week 12
Description: The Mayo Clinic Score is comprised of 4 parts: stool frequency, rectal bleeding, endoscopic findings and physician's global assessment, each scored from 0-3. The total score ranges from 0-12 with higher scores indicating increased severity of disease. Clinical remission is defined as a total Mayo Clinic score of ≤ 2 and no subscores > 1.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | KHK4083 Cohort 1 | KHK4083 Cohort 2 | KHK4083 Cohorts 3 + 4 Combined | KHK4083 Combined | Placebo
Number analyzed (Participants) | 7 | 8 | 22 | 37 | 15
Participants | 1 | 3 | 6 | 10 | 3

13. Secondary Outcome: Number of Subjects Who Achieve Clinical Remission at Week 52
Description: as for outcome 12
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | KHK4083 Cohort 1 | KHK4083 Cohort 2 | KHK4083 Cohorts 3 + 4 Combined | KHK4083 Combined | Placebo
Number analyzed (Participants) | 7 | 8 | 21 | 36 | 14
Participants | 1 | 3 | 6 | 10 | 5

ADVERSE EVENTS:
Time Frame: 52 Weeks
Groups:
- KHK4083 Cohort 1: Subjects who qualify will receive 1.0 mg/kg IV infusion treatments of KHK4083 from Baseline to Week 48.
- KHK4083 Cohort 2: Subjects who qualify will receive 3.0 mg/kg IV infusion treatments of KHK4083 from Baseline to Week 48.
- KHK4083 Cohort 3: Subjects who qualify will receive 10.0 mg/kg IV infusion treatments of KHK4083 from Baseline to Week 48.
- KHK4083 Cohort 4: Subjects who qualify will receive maximum tolerated dose (10.0 mg/kg) IV infusion treatments of KHK4083 from Baseline to Week 48.
- KHK4083 Combined: The total number of participants analyzed who were randomized to KHK4083 during Treatment parts A & B.
Arm/Group | KHK4083 Cohort 1 | KHK4083 Cohort 2 | KHK4083 Cohort 3 | KHK4083 Cohort 4 | KHK4083 Combined | Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 1/10 | 0/9 | 0/21 | 1/49 | 0/17
Serious Adverse Events (participants affected / at risk) | 1/9 | 1/10 | 1/9 | 3/21 | 6/49 | 3/17
Other Adverse Events (participants affected / at risk) | 5/9 | 7/10 | 7/9 | 13/21 | 32/49 | 13/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KHK4083 Cohort 1 (N=9) | KHK4083 Cohort 2 (N=10) | KHK4083 Cohort 3 (N=9) | KHK4083 Cohort 4 (N=21) | KHK4083 Combined (N=49) | Placebo (N=17)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood albumin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abscess drainage (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KHK4083 Cohort 1 (N=9) | KHK4083 Cohort 2 (N=10) | KHK4083 Cohort 3 (N=9) | KHK4083 Cohort 4 (N=21) | KHK4083 Combined (N=49) | Placebo (N=17)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 0 (0) | 3 (3) | 7 (7) | 3 (4)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal aplasia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 5 (5) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Mucous stools (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 6 (6) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scar (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood creatine phosphokinase abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (3) | 1 (1)
Blood folate decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oropharyageal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-10-04): https://cdn.clinicaltrials.gov/large-docs/66/NCT02647866/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-06): https://cdn.clinicaltrials.gov/large-docs/66/NCT02647866/SAP_001.pdf